CLINICAL TRIAL: NCT06119971
Title: Effect of Acupressure on the "Yin-Tang" and "Shen-Men" Points on Pre and Postoperative Anxiety in Elective Caesarean Section: a Prospective, Single-blind, Randomised, Controlled Trial
Acronym: ACUCESAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACUCESAR
Record Dates: First submitted 2023-10-02; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Cesarean Section; Pregnancy; Preoperative Anxiety
Keywords: Acupressure; STAI (State Trait Anxiety Inventory); EDA (Electrodermal Activity)
MeSH Terms: interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: In this study, the acupuncturist is a registered anaesthetist doctor (=investigator) who also holds the Acupuncture Diploma of the Medicine Faculty of Paris. After opening an opaque and sealed envelope, this acupuncturist is in charge of stimulating the true or sham points for each patient, according to the allocated group. As an anaesthetist, he is also responsible of carrying out the anaesthesia. The other care providers (anaesthetic nurses and surgeons) and the patients are blinded. Notably, the primary outcome consists of a self-administered questionnaire. Moreover, to prevent any difference or modification in care according to the results of the questionnaire, the latter is only recovered when the patient leaves the postoperative recovery room. The randomisation list was created with EXCEL software. Finally, an independent person is in charge of the statistical analysis.
  Considering the above, we describe the study as "single-blind".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACUPLUS (Experimental): ACU+ : patients receives stimulation on the true experimental points (Yin-Tang + Shen-Men)
  Interventions: Device: ACUPRESSURE
- ACUMOINS (Placebo Comparator): ACU- : patients receives stimulation on placebo points ("sham" point)
  Interventions: Device: ACUPRESSURE

INTERVENTIONS:
Device: ACUPRESSURE — Acupressure using disposable devices consisting of a metal microbead and an adhesive material.

SUMMARY:
Preoperative anxiety occurs commonly in elective caesarean section and is associated with increased perioperative morbidity. Some groups have used non-pharmacological techniques such as acupressure for its treatment since drugs cross the placenta.

DETAILED DESCRIPTION:
Preoperative anxiety occurs commonly in elective caesarean section and is associated with increased perioperative morbidity. Some groups have used non-pharmacological techniques such as acupressure for its treatment since drugs cross the placenta.

The aim of this study is to examine the efficacy of acupressure with co-stimulation of the "Yin-Tang" and "Shen-Men" points on the reduction in pre- and postoperative anxiety in elective caesarean section.

A single-blind, randomised, controlled, single-centre study will be conducted in ASA I or II patients undergoing elective caesarean section under perispinal anaesthesia. Patients will be randomised into two groups: the ACU+ group (co-stimulation of the "Yin-Tang" and "Shen-Men" points) and the ACU- group (stimulation of two sham points). Anxiety will be assessed using the State-Trait Anxiety Inventory (STAI) score and by measuring skin conductance (Electrodermal Activity [EDA]) during three periods: period 1 (at inclusion, in the patient's hospital room on the morning of the procedure), period 2 (before arrival in the operating theatre) and period 3 (in the postoperative recovery room). True or sham acupressure will be applied using adhesive beads positioned between periods 1 and 2 and left in place until the end of period 3.

ELIGIBILITY:
Inclusion Criteria:

* informed consent obtained
* adult patients
* ASA class I or II
* scheduled caesarean section at CHRU Tours Maternity
* under perispinal anaesthesia (spinal anaesthesia or spinal and epidural anaesthesia combined)

Exclusion Criteria:

* higher or equal to ASA class III
* heart rhythm disorder
* treated with a psychotropic drug (anxiolytic, sedative, antidepressant, antipsychotic, mood stabilizer)
* psychiatric history
* drug or alcohol abuse
* local contraindications to acupuncture (local signs of infection or inflammation, scars)
* scheduled to caesarean section under general anaesthesia.

Patients will be excluded in the event of transition to general anaesthesia or cancellation of the procedure.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
State Trait Anxiety Inventory (STAI) score | At inclusion (the inclusion takes place on the morning of the surgery)
  Difference between the two groups (ACU+ versus ACU-) in STAI score
State Trait Anxiety Inventory (STAI) score | At the entrance in the operative room (this event takes place from 20 minutes to 12 hours after the inclusion, depending on the availability of the surgeons to start the C-section)
  Difference between the two groups (ACU+ versus ACU-) in STAI score
State Trait Anxiety Inventory (STAI) score | In the postoperative recovery room (this event takes place from 40 minutes to 16 hours after the inclusion, depending on the availability fo the surgeons to start the C-section and the duration of this one)
  Difference between the two groups (ACU+ versus ACU-) in STAI score

SECONDARY OUTCOMES:
Electrodermal Activity (EDA) | At inclusion
  Difference between the two groups (ACU+ versus ACU-) in EDA
Electrodermal Activity (EDA) | At the entrance in the operative room (this event takes place from 20 minutes to 12 hours after the inclusion, depending on the availability of the surgeons to start the C-section)
  Difference between the two groups (ACU+ versus ACU-) in EDA
Electrodermal Activity (EDA) | In the postoperative recovery room (this event takes place from 40 minutes to 16 hours after the inclusion, depending on the availability fo the surgeons to start the C-section and the duration of this one)
  Difference between the two groups (ACU+ versus ACU-) in EDA

CONTACTS AND LOCATIONS:
Overall Officials: Marc LAFFON, MD,PhD, Principal Investigator — University Hospital, Tours
Locations (1):
- University Hospital Tours, Tours, France

IPD SHARING:
Plan to Share IPD: No